CLINICAL TRIAL: NCT07102134
Title: The Modified Clipped Ligation of Intersphincteric Fistula Tract (Clipped-LIFT) for High Transsphincteric or Suprasphincteric Fistula: a Proof-of-concept Study
Brief Title: The Modified Clipped-LIFT Procedure for High Transsphincteric or Suprasphincteric Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-053; 1010PY(2023)-03 (Other Grant/Funding Number: Sixth Affiliated Hospital of Sun Yat-Sen University Clinical Research -'1010'Program")
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Anal Fistula Surgery; Anal Fistula
Keywords: High anal fistula; Ligation of the Intersphincteric Fistula Tract procedure; Sphincter-preserving; Clipped ligation.
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suturing-LIFT (Active Comparator): This group received conventional ligation with absorbable sutures
  Interventions: Procedure: Suturing-LIFT procedure
- Clipped-LIFT (Experimental): This group was treated with absorbable clips commonly used for vascular or biliary duct occlusion
  Interventions: Procedure: Clipped-LIFT procedure

INTERVENTIONS:
Procedure: Suturing-LIFT procedure — This group received conventional ligation with absorbable sutures
  Arms: Suturing-LIFT
Procedure: Clipped-LIFT procedure — This group was treated with absorbable clips commonly used for vascular or biliary duct occlusion
  Arms: Clipped-LIFT

SUMMARY:
A retrospective analysis was performed on 96 patients who underwent modified LIFT procedures to treat transsphincteric or suprasphincteric fistulas. Two distinct methods were utilized to ligate the internal sphincter side of the intersphincteric tract: one group received conventional ligation with absorbable sutures (Suturing-LIFT, n=74), while the other group was treated with absorbable clips commonly used for vascular or biliary duct occlusion (Clipped-LIFT, n=22). The primary outcome was the one-stage healing rate, which was compared between the two groups, and the safety profile of the clipped-LIFT approach was analyzed. Both univariate and multivariate analyses were conducted to identify potential prognostic factors associated with therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) preoperative pelvic MRI confirming Parks classification; (2) all patients undergoing a modified LIFT procedure, either with suture ligation (suturing-LIFT group) or clip ligation (clipped-LIFT group).

Exclusion Criteria:

* (1) presence of secondary rectal or anal openings identified as unsuitable for LIFT during postoperative evaluation; (2) lack of clinical outcomes following initial modified LIFT procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
the one-stage healing rate | Complete wound healing without discharge more than 6 months after the modified LIFT procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT07102134/Prot_SAP_000.pdf